CLINICAL TRIAL: NCT05618600
Title: Scripps-eMed Covid-19 Study: A Prospective Monitoring Study for Those Individuals Treated With Paxlovid
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: eMed (Unknown)
Responsible Party: Principal Investigator, Jay Pandit, Study Principal Investigator, Scripps Translational Science Institute
Other Study IDs: ScrippsTSI
Record Dates: First submitted 2022-11-11; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
Keywords: Paxlovid; Rebound; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paxlovid Cohort: Participants will be separated into 2 arms that are self-selected through the decision to opt in or out of Paxlovid. After patients are offered a 5-day course of Paxlovid and have made a treatment decision they will be eligible to join the study. Arm 1 will include 400 participants that opt to take the 5-day course of Paxlovid. Participation will look identical in this study.
- Control Cohort: Participants will be separated into 2 arms that are self-selected through the decision to opt in or out of Paxlovid. After patients are offered a 5-day course of Paxlovid and have made a treatment decision they will be eligible to join the study. Arm 2, control, will include 400 participants that opt out of taking the 5-day course of Paxlovid. Participation will look identical in this study.

SUMMARY:
A prospective monitoring study for those individuals treated with Paxlovid

DETAILED DESCRIPTION:
The purpose of this study is to understand the epidemiology and pathophysiology of Paxlovid rebound in patients with acute Covid-19 infection who have been prescribed the Paxlovid per standard of care.

The study will be a collaborative effort between Scripps and eMed, digitally recruiting 800 participants who have tested positive for Covid-19 and have agreed to be prescribed Paxlovid on the eMed platform.

The vision of the study is to understand Paxlovid rebound and ultimately inform management of acute Covid-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Covid positive
* Qualified for Paxlovid prescription (treatment decision already made prior to enrollment)

Exclusion Criteria:

* Non-english speaking
* Resides outside of the United States

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be obtained from the eMed platform and will consist of participants that tested positive using an eMed rapid antigen test, who underwent a telemedicine visit and opted in or out of receiving a prescription for a 5-day course of Paxlovid.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Paxlovid Rebound | 16 day period
  Incidence of paxlovid rebound defined as test positivity after a documented negative rapid antigen test post 5 day course of Paxlovid

OTHER OUTCOMES:
Symptomatology long term | 6 month period
  Understand the long term impact of paxlovid rebound on symptomatology
Number of viral rebound | 16 day period
  Differences in viral rebound between control and paxlovid group
Number of grouped symptomatology | 16 day period
  Differences in symptomatology between control and paxlovid group.
Immune profile | 6 month period
  Differences in immune profile between control and paxlovid group
Viral Evolution | 6 month period
  Differences in viral evolution between control and paxlovid group

CONTACTS AND LOCATIONS:
Overall Officials: Jay Pandit, MD, Principal Investigator — Scripps Research Institute
Locations (1):
- Scripps Research Institute, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided